CLINICAL TRIAL: NCT06939725
Title: Outcomes of Postoperative Analgesia Protocols and Their Impact on Recovery Quality in Patients Undergoing Cesarean Section
Brief Title: Transverse Abdominis Plane (TAP) Block Versus Transversalis Fascia Plane Block (TFPB) After Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: GOKAEK 2024/22/14
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Acute Pain Management; Caesarean Section
Keywords: ObsQoR-10; Transversalis fascia plane block; Caesarean Section; Transverse abdominis plane block; numeric rating scale
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Transversus abdominis plane block was performed immediately after cesarean section.
  Interventions: Other: Transversus abdominis plane (TAP) block
- Group 2: Transversalis fascial plane block was performed immediately after cesarean section
  Interventions: Other: Transversalis Fascia Plane Block

INTERVENTIONS:
Other: Transversus abdominis plane (TAP) block — We apply different nerve blocks to patients for pain relief after cesarean surgery. Transversus abdominis plane block was applied to this group
  Groups: Group 1
Other: Transversalis Fascia Plane Block — We apply different nerve blocks to patients for pain relief after cesarean surgery. Transversalis Fascia Plane Block was applied to this group
  Groups: Group 2

SUMMARY:
Postoperative analgesia treatment methods are applied to the living in the operating room. It is a routine part of the process of these applications. It is necessary from medical and ethical perspectives. Postoperative analgesia applications are started in the preoperative period and continue in the postoperative period. The analgesic treatment to be used is shaped according to the application and experience of the anesthesiologist. The scientifically accepted developed method is multimodal analgesia protocols. These protocols cover a wide range from paracetamol to opioids, peripheral and central blocks (such as Transversalis Fascial Plane Block (TFPB) and Transversus Abdominis Plane (TAP) Block). The aim of this study is to continue the analgesia protocols applied in cesarean section surgeries on the first 24-hour pain scores, the amount of opioid consumed after surgery and the quality of obstetric recovery (ObsQoR-10) scale.

DETAILED DESCRIPTION:
Postoperative analgesia treatment methods are applied to the living in the operating room. It is a routine part of the process of these applications. It is necessary from medical and ethical perspectives. Postoperative analgesia applications are started in the preoperative period and continue in the postoperative period. The analgesic treatment to be used is shaped according to the application and experience of the anesthesiologist. The scientifically accepted developed method is multimodal analgesia protocols. These protocols cover a wide range from paracetamol to opioids, peripheral and central blocks (such as Transversalis Fascial Plane Block (TFPB) and Transversus Abdominis Plane (TAP) Block). In this study, transversus abdominis plane block or transversalis fascial plane block was applied to the participants immediately after surgery. The aim is to continue the analgesia protocols applied to the cesarean section surgeries on the pain scores in the first 24 hours, the amount of opioid consumed after surgery and the quality of obstetric recovery (ObsQoR-10) scale.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years
2. Term pregnancies (37-42 weeks) and those planned to undergo elective cesarean delivery under spinal anesthesia

Exclusion Criteria:

1. <18 years
2. Emergency surgery
3. BMI > 35 kg/m2 or anatomic conditions that would preclude spinal anesthesia
4. Increased susceptibility to bleeding or coagulation disorders (platelet count below 80,000× 10^3/mm^3 or INR > 1.5)
5. Known allergy to any drug, such as local anesthetics, opioids, or NSAIDs
6. Other relevant maternal or neonatal clinical conditions requiring treatment and at the discretion of the investigators, such as gestational hypertension, impaired renal or hepatic function, postpartum hemorrhage
7. Chronic pain conditions and concomitant use of analgesics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Study Population: Participants who underwent elective cesarean section and received regional anesthesia for postoperative analgesia
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | postoperative 24 hours
  Pain levels of patients will be evaluated with the Numerical Pain Scale (NRS) in the first 24 hours postoperatively.
  The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"

SECONDARY OUTCOMES:
ObsQoR-10 | Postoperative 24 hours
  The ObsQoR-10 questionnaire consists of 10 questions that assess the patient-reported quality of recovery in obstetric patients' postoperative period using an 11-point Likert scale (0 = strongly negative; 10 = strongly positive) that points to a minimum score of 0 (worst possible recovery) and a maximum score of 100 (best possible recovery)

CONTACTS AND LOCATIONS:
Overall Officials: SEVDA AKDENIZ, Assoc Prof, Principal Investigator — Samsun University; HATİCE SELÇUK KUŞDERCİ, Asst. Prof., Study Director — Samsun University
Locations (1):
- Samsun University, Training and Research Hospital, Samsun, İ̇lkadim, Turkey (Türkiye)